CLINICAL TRIAL: NCT01960894
Title: Non-invasive Pressure-Volume Analysis (NIPVA): Extending Comprehensive Left Ventricular Pump Function Assessment to More Patients and Settings
Brief Title: Non-invasive Pressure-Volume Analysis (NIPVA)
Acronym: NIPVA
Status: Completed | Type: Observational
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Other Study IDs: Protocol_NIPVA Study_v1_050613
Record Dates: First submitted 2013-10-09; First posted 2013-10-11 (Estimated); Last update posted 2022-04-11 (Actual); Status verified 2020-01

CONDITIONS: Heart Failure
Keywords: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
If the heart fails to pump a sufficient amount of blood, it is crucial to know why in order to provide the best treatment. Pressure-volume analysis is the gold standard for evaluating the heart's pumping function. Unfortunately, current techniques are invasive, so most patients will not get this examination. By combining the strengths of echo-Doppler ultrasound, blood pressure monitoring and biomedical computing, the investigators aim to develop a non-invasive method for pressure-volume analysis, extending its applicability to more patients and settings.

DETAILED DESCRIPTION:
Background: Current methods to evaluate left ventricular (LV) function either are invasive, precluding routine use in the majority of patients, or fail to discriminate myocardial, hemodynamic and structural factors, rendering assessment imprecise and incomplete.

Key question: Can we reliably obtain LV functional characteristics by non-invasive means, while being able to differentiate more precisely the factors involved? Proposed research: The study team aims to develop a non-invasive method for pressure-volume analysis (NIPVA) of the LV by combining echo-Doppler, peripheral blood pressure measurements and biomechanical modelling. The validity of this approach will be established by comparison with gold standard invasive measurements of pressure-volume relationships in patients undergoing cardiac catheterization. Test-retest reproducibility will be also assessed. The study team hypothesises that NIPVA will provide reproducible and valid measures of LV function and be more widely applicable.

ELIGIBILITY:
Inclusion Criteria:

* Individuals, male or female, aged 18-80 years.
* 30 patients awaiting elective diagnostic coronary angiography will be recruited.
* 30 patients attending cardiology out-patient clinics will be recruited.

Exclusion Criteria:

* Patients with atrial fibrillation or other dysrhythmias or those unable to fully comply with the protocol will be excluded

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients attending cardiology out-patient clinics
Sampling Method: Non-Probability Sample
Enrollment: 65 (Actual)
Dates: Start 2013-10 (Actual); Primary Completion 2016-01 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Reproducibility of non-invasive pressure-volume analysis. | Immediate
  Reproducibility of test-retest non-invasive pressure-volume analysis
Agreement between invasive and non-invasive pressure-volume analysis | Immediate
  Agreement between invasive and non-invasive pressure-volume analysis

CONTACTS AND LOCATIONS:
Overall Officials: Alun Hughes, Principal Investigator — Imperial College London
Locations (1):
- Imperial College Healthcare NHS Trust, Hammersmith Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Heusinkveld MHG, Delhaas T, Lumens J, Huberts W, Spronck B, Hughes AD, Reesink KD. Augmentation index is not a proxy for wave reflection magnitude: mechanistic analysis using a computational model. J Appl Physiol (1985). 2019 Aug 1;127(2):491-500. doi: 10.1152/japplphysiol.00769.2018. Epub 2019 May 30. PMID 31161882